CLINICAL TRIAL: NCT02578433
Title: Mindful Self Compassion in Rehabilitation Inpatients: a Randomized Controlled Trial
Brief Title: Mindful Self Compassion in Rehabilitation Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinik für Psychiatrie und Psychotherapeutische Medizin (Other)
Collaborators: pro mente REHA (Other)
Responsible Party: Principal Investigator, Mag. Lisza Gaiswinkler, Mag. Lisza Gaiswinkler, Universitätsklinik für Psychiatrie und Psychotherapeutische Medizin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECS 1392/2015
Record Dates: First submitted 2015-10-09; First posted 2015-10-19 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Meditation; Progressive Muscle Relaxation
Keywords: Mindful Self Compassion short form; Progressive Muscle Relaxation
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindful Self Compassion (Experimental): Participants will receive a shortened form (6 weeks) of mindful self compassion meditation, once a week for 75 minutes, furthermore they get an audio cd and a handout to practice during the week
  Interventions: Behavioral: Mindful Self Compassion
- Progressive Muscle Relaxation (Other): Participants will receive progressive muscle relaxation once a week for 75 minutes, furthermore they get an audio cd and a handout to practice during the week
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Mindful Self Compassion — Mindful Self Compassion (MSC) training has its primary focus on developing a friendly relationship with oneself by meditation,conversation with the group and the trainer, informal practice and homework assignments. These relationship is founded on mindfulness; therefore the participants will learn a way concentrate on the present moment. The orginal MSC training by Neff and Germer is well established, this intervention will be a shortened form of the original version and will last for the whole visit of the clinical patients in rehabilitation
  Arms: Mindful Self Compassion
Behavioral: Progressive Muscle Relaxation — Progressive Muscle Relaxation by Jacobson is a well known relaxation technique where participants learn to recognize the difference between tension and relaxation by tensing and subsequently relaxing the muscles. The trainingw ill last the wohole stay and the control group will also do homework assignments.
  Arms: Progressive Muscle Relaxation

SUMMARY:
In recent years there has been convincing evidence of the positive effects of mindfulness based interventions, as a form of complementary and alternative medicine in regards to subjective well-being and physical health. There is growing evidence concerning the positive effects of these techniques in regards to an adequate stress management (e.g. respiration and heart rate variability). These findings can be found as well documented in the literature. For this study it is conducted to gain further insights into the role of mindfulness based meditation techniques for psychological well-being. Therefore it is intended to focus on clinical groups (e. g. depression and anxiety patients) in order to find out more about the relevance of mindfulness based meditation techniques as an adjunct for psychiatric and psychotherapeutic treatment. In this study special aspects of mental and spiritual health (e.g. self compassion, subjective perceived stress, spiritual well-being, and psychiatric symptoms) should be examined by comparing a group of clinical patients which practice mindfulness based meditation once a week with a control group, practicing PMR (progressive muscle relaxation)

DETAILED DESCRIPTION:
A holistic view of man is increasingly becoming our consciousness these days. Simultaneously, the demand for efficient and cost-effective forms of treatment for mental illness rises. According to a study by the World Health Organization (2011), 37% of "healthy" working years are lost due to psychiatric disorders. Thus complementary-alternative methods (CAM) as mindfulness-based meditation are becoming more important in medicine. A special form of mindfulness meditation-based training offers "Mindful Self Compassion (MSC)" (to German: achtsames Selbstmitgefühl). As evidence-based sister program to the well-established procedure MBSR and MBCT, MSC provides about meditation, interpersonal exercises, informal practical exercises and homework, the opportunity to learn an attentive and loving contact with itself or to improve and thus contribute effectively to comprehensive well-being. The literature reveals that MSC helps to lead a fulfilling life and is positively related to life satisfaction, emotional intelligence, happiness, optimism and personal initiative. MSC is further negatively correlated with depression, anxiety, self-criticism, the suppression of negative emotions and a negative body image. Furthermore, it is apparent from a study by Blatt (1995) that patients who are very critical towards themselves tend to have less positive effects of antidepressants, placebo and psychotherapy. For this reason it seems of enormous relevance to develop and evaluate therapies, which can help to change people's perception of oneself, like MSC. Based on these results, which show a clear link between Self-Compassion and psychological well-being, a study should be carried out which examines the effects of mindful self compassion meditation on psychological well-being and the severity of clinical symptoms and thus allows a first assessment of effectiveness in clinical practice. A randomized controlled trial is investigated at the rehabilitation center "Sonnenpark Rust Neusiedlersee" where one group of patients (at least 70 patients anticipated) will undergo a shortened form (6 weeks, 75 minutes per week) of MSC training, compared to a group of patients (at least 70 patients anticipated) who undergo regular progressive muscle relaxation (PMR). Both trainings will take place once a week for 6 weeks and will each last for 75 minutes. Patients in both groups will be asked for homework assignments and will get a handout. All relevant parameters are examined at the beginning of the rehabilitation, as well as at the end of the stay at the center. A follow- up after 6 months is planned.

ELIGIBILITY:
Inclusion Criteria:

* Written consent for study participation
* age over 18

Exclusion Criteria:

* psychotic episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Self-Compassion Scale (SCS) | Change from Baseline values in SCS at 6 weeks, follow up 6 months after study completion
  Self compassion is captured via 26 items on a 5-point rating scale. Self Compassion is measured at the beginning and at the end of the 6 weeks intervention

SECONDARY OUTCOMES:
Brief Symptom Inventory (BSI-18) | Change from Baseline values BSI-18 at 6 weeks, follow up 6 months after study completion
  Anxiety, Depression and Somatization as subscales and General Symptom Burden as global score are captured via 18 items on a 4-point rating scale.
Health Survey (SF-36) | Change from Baseline values in SF-36 at 6 weeks, follow up 6 months after study completion
  Health-related quality of life is captured via 36 items over different answering conditions and has 8 subscales: physical functioning, physical role ,bodily pain, general health perceptions, vitality, social functioning, emotional role function and mental well-being

OTHER OUTCOMES:
Sociodemographic Data/ Age | Baseline sociodemographic data, follow up 6 months after study completion
  Digits entry
Sociodemographic Data/ Education | Baseline sociodemographic data, follow up 6 months after study completion
  Education will be assessed by a 6-point rating scale: 1=compulsory education, 2= completed apprenticeship, 3=vocational high school, 4=high school, 5=college degree, 6= university degree and subsequently categorized (1=low education level (compulsory education, completed apprenticeship, vocational high school; 2= high education level (high school, college degree, university degree)
Sociodemographic Data/ Diet | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  Dietary habits will be assessed by a 5-point rating scale (1=with meat, 2=with little meat, 3=with meat and rich in fruits and vegetables, 4=vegetarian with milk/eggs and/or fish, 5=vegan)
Sociodemographic Data/ Weight and Height (BMI) | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  Weight (kg) and Height (m) will be assessed by digits entry and subsequently transformed into BMI
Sociodemographic Data/ Confession | Baseline sociodemographic data, follow up 6 months after study completion
  Confession will be assessed by a 7-point rating scale (1=buddhism, 2=christianity 3=hinduism, 4=islam, 5=judaism, 6=none, 7=other)
Sociodemographic Data/ Diagnosis | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  Diagnosis will be assessed by free answer and subsequently diagnosis will be categorized
Sociodemographic Data/ Medication | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  Medication will be assessed by free answer and subsequently diagnosis will be categorized
Sociodemographic Data/ Level of Perceived Stress | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  Level of Perceived Stress will be captured via 10 point rating scale (1=not at all - 10= absolutely)
Sociodemographic Data/ Previous Experience with Meditation | Baseline sociodemographic data
  dichotomous response format (0=no, 1=yes)
Sociodemographic Data/ Previous Experience with Progressive Muscle Relaxation | Baseline sociodemographic data
  dichotomous response format (0=no, 1=yes)
Sociodemographic Data/ Previous Experience with Mindfulness | Baseline sociodemographic data
  dichotomous response format (0=no, 1=yes)
Sociodemographic Data/ Employment | Baseline sociodemographic data, follow up 6 months after study completion
  Employment will be assessed via 4-point rating scale (1=standing in the Profession, 2=in education, 3=retired, 4=without gainful employment)
Sociodemographic Data/ Marital Status | Baseline sociodemographic data, follow up 6 months after study completion
  Marital Status will be assessed via 4-point rating scale (1=married, 2=partnership, 3=single, 4=widowed/divorced)
Sociodemographic Data/ Alcohol Consumption | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  dichotomous response format (0=no, 1=yes)
Sociodemographic Data/ Drug Consumption | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  dichotomous response format (0=no, 1=yes)
Sociodemographic Data/ Nicotine Consumption | Changes from Baseline sociodemographic data at 6 weeks, follow up 6 months after study completion
  dichotomous response format (0=no, 1=yes), if answered with "yes" it is asked for the amount of cigarettes consumed per day
Sociodemographic Data/ Sympathy of the learned practice (either MSC or PMR) | sociodemographic data at 6 weeks, follow up 6 months after study completion
  will be captured via 10 point rating scale (1=not at all - 10= absolutely)
Sociodemographic Data/ Sympathy of the trainer (either MSC or PMR) | sociodemographic data at 6 weeks, follow up 6 months after study completion
  will be captured via 10 point rating scale (1=not at all - 10= absolutely)
Sociodemographic Data/ Duration of Practice | sociodemographic data at 6 weeks, follow up 6 months after study completion
  dichotomous response format (0=no, 1=yes), if answered with "yes" (I practice MSC/PMR) it is asked for the amount of practice per day with a 3-point rating scale (1=less than 10 minutes, 2= 10-15 minutes, 3=more than 15 minutes)
Sociodemographic Data/ Frequency of Practice | sociodemographic data at 6 weeks, follow up 6 months after study completion
  dichotomous response format (0=no, 1=yes), if answered with "yes" (I practice MSC/PMR) it is asked for the frequency of practice per day with a 4-point rating scale (1=daily, 2=serveral times a week, 3=once per week, 4=less than once a week)
Sociodemographic Data/ Type of Practice | sociodemographic data at 6 weeks, follow up 6 months after study completion
  dichotomous response format (0=no, 1=yes), if answered with "yes" (I practice MSC/PMR) it is asked for the type (ritualized vs. informal) of practice
Subjective Feeling of Health | Changes from Baseline data at 6 weeks, follow up 6 months after study completion
  will be captured via 10 point rating scale (1=not at all - 10= absolutely)
Subjective Feeling of Happines | Changes from Baseline data at 6 weeks, follow up 6 months after study completion
  will be captured via 10 point rating scale (1=not at all - 10= absolutely)
Previous Experience with Yoga | Baseline sociodemographic data, captured at the beginning
  dichotomous response format (0=no, 1=yes)
Previous Experience with Mindful Self Compassion | Baseline sociodemographic data, captured at the beginning
  dichotomous response format (0=no, 1=yes)

CONTACTS AND LOCATIONS:
Overall Officials: Human-Friedrich Unterrainer, Priv.Doz., Principal Investigator — Universitätsklinik für Psychiatrie/Medizinische Univeristät Graz
Locations (1):
- Universitätsklinik für Psychiatrie und Psychotherapeutische Medizin, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balasubramaniam M, Telles S, Doraiswamy PM. Yoga on our minds: a systematic review of yoga for neuropsychiatric disorders. Front Psychiatry. 2013 Jan 25;3:117. doi: 10.3389/fpsyt.2012.00117. eCollection 2012. PMID 23355825
- [Background] Barnett JE, Shale AJ. The Integration of Complementary and Alternative Medicine (CAM) into the Practice of Psychology: A Vision for the Future. Professional Psychology. Resarch and Practice 43: 576-585, 2012.
- [Background] Foryflow AL. Integrating Yoga with Psychotherapy: A Complementary Treatment for Anxiety and Depression. Canadian Journal of Counselling and Psychotherapy 45: 132-150, 2011.
- [Background] World Health Organization. Global Status Report on Non-Communicable Diseases. Geneva:WHO 2010, 2011.
- [Background] Blatt SJ. Representational structures in psychopathology. University of Rochester Press 6: 1-34, 1995
- [Background] Bullinger M. German translation and psychometric testing of the SF-36 Health Survey: preliminary results from the IQOLA Project. International Quality of Life Assessment. Soc Sci Med. 1995 Nov;41(10):1359-66. doi: 10.1016/0277-9536(95)00115-n. PMID 8560303
- [Result] Spitzer C, Hammer S, Lowe B, Grabe HJ, Barnow S, Rose M, Wingenfeld K, Freyberger HJ, Franke GH. [The short version of the Brief Symptom Inventory (BSI -18): preliminary psychometric properties of the German translation]. Fortschr Neurol Psychiatr. 2011 Sep;79(9):517-23. doi: 10.1055/s-0031-1281602. Epub 2011 Aug 25. German. PMID 21870312
- [Result] Neff KD. Development and validation of a scale to measure self-compassion. Self and Identity 2: 223-250, 1993.